CLINICAL TRIAL: NCT07288658
Title: Comparing the Fit and Performance of Scleral Lenses With Oval and Circular Limbal Zones
Acronym: CHIMERA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Fighting Blindness Canada (Unknown); Canadian Optometric Education Trust Fund (COETF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 47580
Record Dates: First submitted 2025-09-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Limbus Corneae
Keywords: limbus; scleral lens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scleral lenses with an oval limbal zone (Experimental): Scleral lenses with an oval limbal zone designed with a scleral lens custom design software (WAVE Contact Lens System)
  Interventions: Device: Scleral lenses
- Scleral lenses with a circular limbal zone (Active Comparator): Scleral lenses with a circular limbal zone designed with a scleral lens custom design software (WAVE Contact Lens System)
  Interventions: Device: Scleral lenses

INTERVENTIONS:
Device: Scleral lenses — Scleral lenses designed with oval and circular limbal zone designs

SUMMARY:
Scleral lenses are large, rigid contact lenses that rest on the white part of the eye and arch over the cornea. They are commonly used to improve vision in people with eye conditions like keratoconus or corneal scarring, but are increasingly popular among people with high prescriptions or dry eyes due to the comfort and clarity they provide.

While these lenses offer many benefits, fitting them properly can be difficult, especially over the limbus, the border between the clear front surface of the eye and the white part of the eye. This area is home to important stem cells that help keep the eye healthy. Most lenses today are designed to fit the limbus as if it were perfectly round, but new research shows the limbus is actually more oval-shaped. When scleral lenses do not match this shape, they may press too hard in some areas or leave too much space in other areas of the limbus, potentially causing discomfort or long-term eye health problems.

This study will test whether lenses designed with an oval-shaped limbal zone provide a better fit and greater comfort than traditional round designs. To do this, advanced eye imaging and computer modelling will be used to measure the limbus and customize scleral lens design for each participant.

All lenses used in the study are already approved and available in Canada. The results may help improve lens comfort and safety for people who rely on scleral lenses every day.

DETAILED DESCRIPTION:
Scleral lenses are large diameter rigid contact lenses with a wide range of clinical applications. Traditionally, scleral lenses are used for visual rehabilitation of patients with irregular corneas, such as patients with keratoconus or corneal scarring. In these patients, scleral lenses are the mainstay of treatment, as they significantly improve visual acuity and quality. Recently, scleral lenses have gained popularity amongst patients without corneal abnormalities for their ability to correct high prescriptions and provide relief from dry eye symptoms. Scleral lenses are a growing field of interest in eye care, and many new technologies have emerged in recent years to assist with scleral lens fitting.

Fitting scleral lenses, however, is not without challenges, and currently available scleral lens fitting strategies may not be adequate for the long-term needs of all patients. In particular, fitting of scleral lenses over the limbal area is known to be suboptimal. The limbus is the transitional area between the clear cornea and the white sclera. It contains numerous limbal stem cells crucial to maintaining long-term corneal health. Currently, the majority of contemporary scleral lens designs only involve a uniform circular-shaped area to fit over the limbus. However, several reports have recently shown that the human limbus is of an oval rather than a circular shape. Furthermore, there is currently limited information on the elevation/height of the limbal zone, including whether the height of the limbal zone is the same or different in each quadrant and whether this should be compensated for in lens design and fitting. The mismatch between the limbal zone design in a scleral lens and the true limbal shape leads to inappropriate fit of scleral lenses in the limbal area: typically, there can be excessive and inadequate clearance over the limbus in different parts of the same eye. Excessive and inadequate clearance both cause stress to the limbal stem cells, which is hypothesized to compromise patient comfort and risk the health of the cornea long-term.

To enhance lens comfort and minimize the risk of compromising ocular health, scleral lenses must be designed with an accurate understanding of the limbus's shape and dimensions. Achieving this requires a reliable and efficient method for capturing and analyzing limbal data. One such method involves a computational approach that uses Zernike polynomial-based modeling to identify limbal points on a corneoscleral topography scan, a technique previously validated on model eye scans. The proposed study will evaluate the performance of scleral lenses with oval versus circular limbal zones, using limbal width measurements obtained through a customized MATLAB program based on this method. The hypothesis is that when compared to scleral lenses designed with a standard, circular, non-customized limbal zone, scleral lenses with an oval limbal zone may result in more even limbal clearance 360, which leads to less corneal observations (e.g. corneal staining, corneal microcysts) related to scleral lens fit issues in the limbal area (e.g. limbal congestion, limbal touch, conjunctival prolapse), less lens decentration and better subjective comfort when worn.

The study lenses are marketed and commercially available in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age and has full legal capacity to volunteer;
* Have signed an information consent letter;
* Are willing and able to follow instructions and maintain the appointment schedule;
* Are existing wearers of WAVE ScleraLens in one or both eyes.

Exclusion Criteria:

* Are participating in any concurrent clinical or research study;
* Have any known active* ocular disease and/or infection;
* Have known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Have taken part in another (pharmaceutical) research study within the last 30 days; * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and mild dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Limbal clearance in 4 semi-meridians (superior, nasal, inferior and temporal) of a scleral lens | at the Follow-up Visits 2 weeks and 4 weeks after the start of the study
  Measured in microns on an Anterion anterior segment OCT scan using the built-in calipers.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — University of Waterloo
Locations (1):
- School of Optometry & Vision Science, University of Waterloo, Waterloo, Ontario, Canada